CLINICAL TRIAL: NCT03403127
Title: Prospective Study of CT and PET Imaging During a Course of Radical Radiotherapy to Determine the Dosimetric Benefits of Re-Planning in Non-Small Cell Lung Cancer
Brief Title: PET CT Re-Planning NSCLC (4DCT-PET)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-0269
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT Scans — PET Imaging requires the use of an investigational drug, a radioactively-labelled sugar called 18F-Fluorodeoxyglucose (FDG). FDG is glucose labelled with a radioactive fluorine atom. It is given by intravenous injection and is particularly absorbed by cancer cells. The radioactive signal given off by the FDG can then be detected by the PET scanner providing an image of the cancer (or tumour).

SUMMARY:
This study will see whether the addition of more frequent planning CTs during the course of radiation, and of Positron Emission Tomography (PET), a diagnostic test similar to CT, prior to and during a course of radiation may provide information that could potentially be used during the treatment to improve the initial radiation plan.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or more than 18 years old
* Patients with NSCLC consenting for radiotherapy to the primary tumor and / or mediastinal / hilar lymph nodes. Prescription doses should be 60Gy or higher.
* Chemo-RT patients of any stage of NSCLC
* Patients with a measurable tumor on CT scan.
* Patients who are able to lie supine for two consecutive 25 minutes sessions.

Exclusion Criteria:

* Trimodality patients who will have surgery within 2 months post RT
* Previous radiotherapy to intended treatment volumes.
* Patients with recurrent disease
* Active malignancy other than lung cancer
* Pregnancy
* Failure to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-05-20 (Actual); Primary Completion 2013-03-25 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
GTV volumes | 2 weeks post RT treatment
  The ratio of the GTV volumes defined using 4D CT (GTV4DCT) planning scans is a prognostic parameter for NSCLC.
GTV volumes | 4 weeks post RT Treatment
  The ratio of the GTV volumes defined using 4D CT (GTV4DCT) planning scans is a prognostic parameter for NSCLC
GTV volumes | 7 weeks post RT Treatment
  The ratio of the GTV volumes defined using 4D CT (GTV4DCT) planning scans is a prognostic parameter for NSCLC
GTV volumes | 3 months post RT treatment
  he ratio of the GTV volumes defined using 4D CT (GTV4DCT) planning scans is a prognostic parameter for NSCLC
GTV volumes | 2 weeks post RT Treatment
  The ratio of the GTV volumes defined using FDG PET (GTVPET) planning scans
GTV Volumes | 4 weeks post RT Treatment
  The ratio of the GTV volumes defined using FDG PET (GTVPET) planning scans
GTV Volumes | 7 weeks post RT Treatment
  The ratio of the GTV volumes defined using FDG PET (GTVPET) planning scans
GTV volumes | 3 months post RT treatment
  The ratio of the GTV volumes defined using FDG PET (GTVPET) planning scans

IPD SHARING:
Plan to Share IPD: Undecided